CLINICAL TRIAL: NCT02567045
Title: Uptake to Colorectal Cancer Screening in Familiar-risk Population: A Randomized Controlled Trial Comparing Immunochemical Fecal Occult Blood Test With Colonoscopy
Brief Title: Uptake to Colorectal Cancer Screening in Familial-risk Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario de Canarias (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Colorectal cancer screening
Record Dates: First submitted 2015-09-29; First posted 2015-10-02 (Estimated); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Colorectal Cancer; Screening Uptake of Colonoscopy and FIT
Keywords: Immunochemical fecal occult blood test; Colonoscopy; Screening uptake; Screening participation; Familiar risk; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Masking Description: Participants were randomized to either colonoscopy or faecal occult blood test
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fecal occult blood testing (Experimental): Annual FIT and colonoscopy in case of a positive test. Fecal occult blood testing: annual FIT (two rounds) without diet restriction, one stool sample. Positive cut-off = 10 μg Hemoglobin/g feces.
  Colonoscopy will be performed in case of a positive FIT.
  Interventions: Procedure: annual FIT and colonoscopy in case of a positive test; Procedure: colonoscopy with sedation
- one-time Colonoscopy (Active Comparator): One-time Colonoscopy with sedation
  Interventions: Procedure: colonoscopy with sedation

INTERVENTIONS:
Procedure: annual FIT and colonoscopy in case of a positive test — FIT and colonoscopy in case of a positive test. Annual interval (2 rounds), without diet restriction, 1 stool sample. Positive cut-off 10 mcg Hemoglobin/g feces.
  Arms: Fecal occult blood testing
Procedure: colonoscopy with sedation — One-time Colonoscopy with sedation.

SUMMARY:
This is a multicenter, controlled, randomized phase III study to compare participation rate with two screening rounds of fecal occult blood test (FIT) versus one-time screening colonoscopy in first degree relatives (FDR) of patients diagnosed of colorectal cancer (CRC).

The hypothesis of the study is that annual FIT uptake and colonoscopy when a positive test is higher than that of straightforward colonoscopy. Assuming an uptake of 0.50 for colonoscopy and 0.60 for FIT, a Type I error (alpha) of 5% and a power of 90%, 538 FDRs will be necessary to include in each group.

DETAILED DESCRIPTION:
This is a multicenter, controlled, randomized phase III study to compare participation rate with two screening rounds of FIT versus one-time screening colonoscopy in FDR of patients diagnosed of CRC.

The recruitment process will be programmed through the index case, that will be interviewed to obtain their CRC family history. FDR will be contacted in order to make an appointment in the High-risk CRC Clinic of the participant centers. Randomization will be performed before signing the informed consent to avoid selection bias. A researcher will be responsible to provide detailed information about the study and getting the informed consent. In case of willingness to participate in the study, the FDR will be randomized to one of the following arms: A) One-time colonoscopy; B) annual FIT for two screening rounds and a colonoscopy in case of a positive FIT (cut-off = 10 μg Hemoglobin/g feces). Screening uptake will be defined as the percentage of FDR who participate at least in one of the two FIT screening round in the FIT group or who undergo colonoscopy in the other group. Screening uptake will be calculated under the assumption of intention to screen analysis.

The hypothesis of the study is that annual FIT uptake and colonoscopy when a positive test is higher than that of straightforward colonoscopy. Assuming an uptake of 0.50 for colonoscopy and 0.60 for FIT, a Type I error (alpha) of 5% and a power of 90%, 538 FDRs will be necessary to include in each group.

ELIGIBILITY:
Inclusion Criteria:

1. FDR with a case index meeting the following conditions: at least one case index < 60 years at diagnosis of the CCR;
2. having ≥ 2 FDRs with CRC regardless the age of the case index at diagnosis;
3. having a sibling with CRC;
4. age <75 years.

Exclusion Criteria:

1. past CRC screening;
2. inflammatory bowel disease or past history of colorectal neoplasia;
3. Family history of hereditary CRC;
4. Abdominal symptoms;
5. Colectomy;
6. Severe comorbidity leading to a poor prognosis (life expectancy < 5 years);
7. Refusal to participate in the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 260 (Actual)
Dates: Start 2016-02-25 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who participate in each screening arm | 2 years

SECONDARY OUTCOMES:
Efficacy measure: QALYs (Quality adjusted life years). | 2 years
Costs measure: cost (euros) of the procedures associated with each screening strategy and treatment of advanced neoplastic lesions | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Quintero, MD, PhD, Study Director — Hospital Universitario de Canarias
Locations (7):
- Spain (7):
  - Federico Sopeña Biarge, Zaragoza, Aragon
  - Cristina Alvarez Urturi, MD, Barcelona, Catalonia
  - Maria Teresa Ocaña Bombardo, Barcelona, Catalonia
  - Inés Castro Novo, Ourense, Galicia
  - Patricia Muñoz Garrrido, San Sebastián, País Vasco, Gipuzcoa
  - Digestive Service, Huc, San Cristóbal de La Laguna, S/C de Tenerife
  - María Rodriguez Soler, Alicante

REFERENCES:
- [Result] Quintero E, Carrillo M, Gimeno-Garcia AZ, Hernandez-Guerra M, Nicolas-Perez D, Alonso-Abreu I, Diez-Fuentes ML, Abraira V. Equivalency of fecal immunochemical tests and colonoscopy in familial colorectal cancer screening. Gastroenterology. 2014 Nov;147(5):1021-30.e1; quiz e16-7. doi: 10.1053/j.gastro.2014.08.004. Epub 2014 Aug 13. PMID 25127679
- [Result] Quintero E, Castells A, Bujanda L, Cubiella J, Salas D, Lanas A, Andreu M, Carballo F, Morillas JD, Hernandez C, Jover R, Montalvo I, Arenas J, Laredo E, Hernandez V, Iglesias F, Cid E, Zubizarreta R, Sala T, Ponce M, Andres M, Teruel G, Peris A, Roncales MP, Polo-Tomas M, Bessa X, Ferrer-Armengou O, Grau J, Serradesanferm A, Ono A, Cruzado J, Perez-Riquelme F, Alonso-Abreu I, de la Vega-Prieto M, Reyes-Melian JM, Cacho G, Diaz-Tasende J, Herreros-de-Tejada A, Poves C, Santander C, Gonzalez-Navarro A; COLONPREV Study Investigators. Colonoscopy versus fecal immunochemical testing in colorectal-cancer screening. N Engl J Med. 2012 Feb 23;366(8):697-706. doi: 10.1056/NEJMoa1108895. PMID 22356323
- [Result] Pappadopulos E, Jensen PS, Chait AR, Arnold LE, Swanson JM, Greenhill LL, Hechtman L, Chuang S, Wells KC, Pelham W, Cooper T, Elliott G, Newcorn JH. Medication adherence in the MTA: saliva methylphenidate samples versus parent report and mediating effect of concomitant behavioral treatment. J Am Acad Child Adolesc Psychiatry. 2009 May;48(5):501-510. doi: 10.1097/CHI.0b013e31819c23ed. PMID 19307987
- [Result] Dove-Edwin I, Sasieni P, Adams J, Thomas HJ. Prevention of colorectal cancer by colonoscopic surveillance in individuals with a family history of colorectal cancer: 16 year, prospective, follow-up study. BMJ. 2005 Nov 5;331(7524):1047. doi: 10.1136/bmj.38606.794560.EB. Epub 2005 Oct 21. PMID 16243849
- [Derived] Gonzalez-Lopez N, Quintero E, Gimeno-Garcia AZ, Bujanda L, Banales J, Cubiella J, Salve-Bouzo M, Herrero-Rivas JM, Cid-Delgado E, Alvarez-Sanchez V, Ledo-Rodriguez A, de-Castro-Parga ML, Fernandez-Poceiro R, Sanroman-Alvarez L, Santiago-Garcia J, Herreros-de-Tejada A, Ocana-Bombardo T, Balaguer F, Rodriguez-Soler M, Jover R, Ponce M, Alvarez-Urturi C, Bessa X, Roncales MP, Sopena F, Lanas A, Nicolas-Perez D, Adrian-de-Ganzo Z, Carrillo-Palau M, Gonzalez-Davila E; Oncology Group of Asociacion Espanola de Gastroenterologia. Screening uptake of colonoscopy versus fecal immunochemical testing in first-degree relatives of patients with non-syndromic colorectal cancer: A multicenter, open-label, parallel-group, randomized trial (ParCoFit study). PLoS Med. 2023 Oct 24;20(10):e1004298. doi: 10.1371/journal.pmed.1004298. eCollection 2023 Oct. PMID 37874831